CLINICAL TRIAL: NCT03467672
Title: Interest of Eosinopia in the Diagnosis of Infection in the Emergency Department
Acronym: SEPSISEO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6228
Record Dates: First submitted 2018-02-12; First posted 2018-03-16 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Eosinopenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infected patients
  Interventions: Other: Diagnosis of bacterial infection
- Control group
  Interventions: Other: Diagnosis of bacterial infection

INTERVENTIONS:
Other: Diagnosis of bacterial infection — use of eosinopenia in the diagnosis of bacterial infection

SUMMARY:
Several studies have described the interest of eosinopenia as a marker of infection in internal medicine or in intensive care units. Eosinopenia is an inexpensive and easily accessible biological marker of sepsis. Retrospective work in the adult emergency departments of Strasbourg University Hospitals has shown the good specificity of this biological sign for the diagnosis of infection. Our work aims to confirm the results by a more meaningful study.

Main objective: Evaluation of the interest of eosinopenia in the diagnosis of bacterial infection in ED.

Methodology: inclusion of all patients with criteria for bacterial infection in ED, inclusion of an equivalent number of uninfected control patients.

Duration : 12 months Multicentric prospective study 6 centers : Strasbourg, Hôpital Nord Franche comté, Sélestat, Wissembourg, Colmar, Mulhouse

ELIGIBILITY:
Inclusion Criteria:

* major patient
* patient suspected of infection and benefiting from the routine practice of NFS, whatever the indication during his / her visit to the emergency room.
* patient with or without criteria for bacterial infection
* patient affiliated to a social security scheme
* patient (or legal representative) who has agreed to participate in the study

Exclusion Criteria:

* anti tumor chemotherapy
* immunosuppressive treatment
* corticotherapy
* antibiotherapy in progress
* malignant hemopathy
* evolutionary cancer
* refusal to participate in the study
* subjects under safeguard of justice
* subject under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult emergency counseling subjects who benefit from the routine practice of NFS for any indication.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
eosinopenia as a sepsis marker | 102 month
  Evaluation of the interest of eosinopenia in the diagnosis of infectious states in emergencies.

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CH de COLMAR, Colmar
  - CH de MULHOUSE, Mulhouse
  - Ch Selestat, Sélestat
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg
  - CH Nord Franche comte, Trévenans
  - Ch Wissembourg, Wissembourg

IPD SHARING:
Plan to Share IPD: Undecided